CLINICAL TRIAL: NCT03414671
Title: The Effect of Standardizing the Definition and Approach to a Clinically Significant Cardiopulmonary Event in Infants Less Than 30 Weeks on Length of Stay
Brief Title: The Effect of Standardizing the Definition of a Clinically Significant Cardiopulmonary Event on Length of Stay
Acronym: CSCPE
Status: Completed | Type: Observational
Sponsor: Pediatrix (Other)
Responsible Party: Sponsor
Other Study IDs: 5892S-15
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Apnea of Prematurity
Keywords: apnea
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- historical control: All infants born < 30 weeks gestation admitted to the Swedish Hospital NICU from 11/30/2015-11/30/2017 (historical control, pre-standardized defined CSCPE
- Standardized: All infants born < 30 weeks gestation admitted to the Swedish Hospital NICU from 6/1/2018 - 12/31/20 (the group following implementation of the standardized defined CSCPE)

SUMMARY:
A health care initiative will be implemented December 4, 2017 in the Newborn Intensive Care (NICU) setting in an attempt to reduce the length of stay (LOS) for premature infants after standardizing the definition and approach to a clinically significant cardiopulmonary event (CSCPE). We would like to compare LOS in infants born < 30 weeks gestation before and after standardization to see if LOS is reduced.

DETAILED DESCRIPTION:
The LOS of infants born < 30 weeks prior to implementation of the standardized definition of a CSCPE (11/30/2015-11/30/2017) will be compared to the LOS for all infants who meet the inclusion criteria and born < 30 weeks from 6/1/2018 - 12/31/20. Data collection will begin June 1,2018, seven months after implementing the CSCPE definition. This will allow time for the nursing staff, the physicians and nurse practitioners to become familiar with the new CSCPE definition and management.

Following implementation of the new definition, the researchers will also do a 6 month audit on nursing response to a CSCPE based on the current alarm settings. Initially we do not plan to change the alarm limits but we may find the lower alarm limits for heart rate and oxygen saturation are set too high and may need to be lowered to more accurately assist nurses in recognizing when an infant is having a CSCPE. If the 6 month audit shows nurses are "missing" a CSCPE because the current lower alarm limits are set too high, or stimulating an infant inappropriately too early, the alarm limits will be changed at every bedside. If the alarm limits are reset, data collection will begin 6 months after the alarms are changed. This is expected to be starting 1/1/2019 and conclude 12/31/20. If it is decided the lower alarm limits will not need to be changed, data collection will begin 6/1/2018 and conclude 8/31/20 instead of 12/31/20.

ELIGIBILITY:
Inclusion Criteria:

* All infants born < 30 weeks gestation admitted to the Swedish Hospital NICU from 11/30/2015-11/30/2017 (historical control, pre-standardized defined CSCPE) and 6/1/2018 - 12/31/20 (the group following implementation of the standardized defined CSCPE).

Exclusion Criteria:

* Those babies who:
* expired during the evaluation periods
* transferred in after 30 weeks PMA
* transferred out and then lost to follow-up
* had a significant congenital, neurological, facial or airway anomaly affecting the infant's breathing beyond 36 weeks PCA
* subjects who are not yet adults (infants, children, teenagers)

Ages: 23 Weeks to 29 Weeks | Sex: All
Age Groups: Child
Study Population: This study will only enroll infants admitted to the Swedish Medical Center First Hill
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-21 (Actual)

PRIMARY OUTCOMES:
LOS - CSCPE | 24 months
  reduce the length of stay (LOS) for premature infants after standardizing the definition and approach to a clinically significant cardiopulmonary event

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kamitsuka, MD, Principal Investigator — Pediatrix
Locations (1):
- Swedish Medical Center First Hill, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barrington KJ, Finer N, Li D. Predischarge respiratory recordings in very low birth weight newborn infants. J Pediatr. 1996 Dec;129(6):934-40. doi: 10.1016/s0022-3476(96)70044-6. PMID 8969742
- [Background] Cote A, Hum C, Brouillette RT, Themens M. Frequency and timing of recurrent events in infants using home cardiorespiratory monitors. J Pediatr. 1998 May;132(5):783-9. doi: 10.1016/s0022-3476(98)70304-x. PMID 9602186
- [Background] Ramanathan R, Corwin MJ, Hunt CE, Lister G, Tinsley LR, Baird T, Silvestri JM, Crowell DH, Hufford D, Martin RJ, Neuman MR, Weese-Mayer DE, Cupples LA, Peucker M, Willinger M, Keens TG; Collaborative Home Infant Monitoring Evaluation (CHIME) Study Group. Cardiorespiratory events recorded on home monitors: Comparison of healthy infants with those at increased risk for SIDS. JAMA. 2001 May 2;285(17):2199-207. doi: 10.1001/jama.285.17.2199. PMID 11325321
- [Background] Jobe AH. What do home monitors contribute to the SIDS problem? JAMA. 2001 May 2;285(17):2244-5. doi: 10.1001/jama.285.17.2244. No abstract available. PMID 11325327
- [Background] Eichenwald EC; Committee on Fetus and Newborn, American Academy of Pediatrics. Apnea of Prematurity. Pediatrics. 2016 Jan;137(1). doi: 10.1542/peds.2015-3757. Epub 2015 Dec 1. PMID 26628729
- [Background] Poets CF, Roberts RS, Schmidt B, Whyte RK, Asztalos EV, Bader D, Bairam A, Moddemann D, Peliowski A, Rabi Y, Solimano A, Nelson H; Canadian Oxygen Trial Investigators. Association Between Intermittent Hypoxemia or Bradycardia and Late Death or Disability in Extremely Preterm Infants. JAMA. 2015 Aug 11;314(6):595-603. doi: 10.1001/jama.2015.8841. PMID 26262797
- [Background] Poets CF, Stebbens VA, Richard D, Southall DP. Prolonged episodes of hypoxemia in preterm infants undetectable by cardiorespiratory monitors. Pediatrics. 1995 Jun;95(6):860-3. PMID 7761210
- [Background] Martin RJ, Wang K, Koroglu O, Di Fiore J, Kc P. Intermittent hypoxic episodes in preterm infants: do they matter? Neonatology. 2011;100(3):303-10. doi: 10.1159/000329922. Epub 2011 Oct 3. PMID 21986336
- [Background] Butler TJ, Firestone KS, Grow JL, Kantak AD. Standardizing documentation and the clinical approach to apnea of prematurity reduces length of stay, improves staff satisfaction, and decreases hospital cost. Jt Comm J Qual Patient Saf. 2014 Jun;40(6):263-9. doi: 10.1016/s1553-7250(14)40035-7. PMID 25016674
- [Background] Adamsons K, Myers RE. Late decelerations and brain tolerance of the fetal monkey to intrapartum asphyxia. Am J Obstet Gynecol. 1977 Aug 15;128(8):893-900. doi: 10.1016/0002-9378(77)90059-x. PMID 407796
- [Background] Juul SE, Aylward E, Richards T, McPherson RJ, Kuratani J, Burbacher TM. Prenatal cord clamping in newborn Macaca nemestrina: a model of perinatal asphyxia. Dev Neurosci. 2007;29(4-5):311-20. doi: 10.1159/000105472. PMID 17762199